CLINICAL TRIAL: NCT01479075
Title: The Effect of Central Insulin on Insulin Sensitivity and Energy Metabolism
Acronym: Centrin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Centrin
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Diabetes
Keywords: central insulin; insulin resistance; energy metabolism
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- intranasal insulin in patients (Experimental): intranasal insulin is applied to diabetic patients under fasting conditions
  Interventions: Drug: intransal insulin
- intransal insulin in study participants (Experimental): intranasal insulin is applied to healthy patients under fasting conditions
  Interventions: Drug: intransal insulin
- placebo in patients (Placebo Comparator): placebo spray is applied intranasally in type 2 diabetes patients under fasting conditions
  Interventions: Drug: Placebo
- placebo in study participants (Experimental): placebo spray is applied intranasally in healthy participants under fasting conditions
  Interventions: Drug: Placebo
- taNVS (Experimental): Transcutanoues auricular vagus nerve stimulation is applied for 14 min in the external ear in healthy participants
  Interventions: Device: taVNS
- Sham stimulation (Placebo Comparator): Sham stimulation in the ear lobe is applied for 14 min in healthy participants
  Interventions: Device: sham stimulation

INTERVENTIONS:
Drug: intransal insulin — 4x 40mU intranasal insulin
  Other Names: intranasal insulin
  Arms: intranasal insulin in patients; intransal insulin in study participants
Drug: Placebo
  Other Names: intranasal placebo spray
  Arms: placebo in patients; placebo in study participants
Device: taVNS
  Other Names: transcutaneous auricular vagus nerve stimulation
  Arms: taNVS
Device: sham stimulation
  Other Names: sham stimulation in the ear lobe
  Arms: Sham stimulation

SUMMARY:
Insulin has a direct effect on the energy metabolism of the brain under basal conditions and has an effect on the hepatic glucose production, lipid metabolism and the secretion of various hormone. The effect of intranasal insulin on peripheral metabolism in humans supposedly is mediated by the vagus nerve.

The purpose of this study is to determine whether central insulin influences the human peripheral insulin sensitivity of liver and muscle and whether vagus nerve stimulation can mimick this effect.

DETAILED DESCRIPTION:
Insulin has a direct effect on the energy metabolism of the brain under basal conditions and has an effect on the hepatic glucose production, lipid metabolism in the mouse model.

The purpose of this study is to determine whether central insulin influences the human peripheral insulin sensitivity of liver and muscle and energy metabolism. Intranasal insulin can be used in humans to deliver insulin to the brain and studies have shown that intranasal insulin might reduce food intake, lower body weight and modulate muscle glucose and adipose tissue lipid metabolism in himans. These effects are likely mediated by the vagus nerve as skeletal muscle insulin sensitization after intranasal insulin relates to parasympathetic tone activity (Heni et al. Diabetes 2014). Transcutaneous auricular vagus nerve stimulation (taVNS) activates non-invasively the sensory branches of the vagus nerve and is applied in humans as adjuvant treatment in drug-resistant epilepsy (Frangos et al. 2015). Thereby it can be used to examine whether the vagus nerve indeed mediates brain insulin signals to the periphery.

Here we aim to investigate the effects of intranasal insulin on hepatic glucose, lipid and energy metabolism. We further aim to test whether taVNS can mimick intranasal insulin effects on peripheral metabolism in humans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 and ≤ 70 years
* balanced gender ratio (50: 50)
* BMI 20-25 kg/m² (normal weight subjects)
* BMI 25-35 kg/m² (obese subjects)

Exclusion Criteria:

* acute illness within the last 2 weeks before the examination
* autoimmune diseases and disorders immune- compromised (leukocytes <5000/μl)
* renal insufficiency (creatinine> 1.5 mg / dl)
* heart disease, condition after heart attack
* anemia (Hb <12 g / l, controls at each examination), blood donation within 4 weeks before the examination
* participation in another study within 2 months before the examination
* wear a metal or magnetic objects on or in the body
* claustrophobia
* use of immunomodulatory drugs (cortisol, antihistamines, aspirin)
* thyroid disease
* taking glitazones and insulin therapy
* pregnancy, lactation, menstruation
* cigarette smoking, use of alcohol or drugs, psychiatric disorders
* risk for / or manifest AIDS (HIV) or hepatitis B or C
* liver disease is not attributed to the existence of a non-alcoholic steatosis
* night shift work or circumstances, which do not allow the normal day-night rhythm
* bleeding disorders or disorders in wound healing
* hypersensitivity to local anesthetics
* malignant cancer
* heart rhythm disorders
* polyneuropathy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 6 months
  Assessment of insulin sensitivity with gold standard methods

SECONDARY OUTCOMES:
Energy metabolism | 6 months
  Energy metabolism is assessed from gold standard methods

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, MD, Prof, Study Director — Germyn Diabetic Center; Julia Szendrödi, MD, PhD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetic Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Frangos E, Ellrich J, Komisaruk BR. Non-invasive Access to the Vagus Nerve Central Projections via Electrical Stimulation of the External Ear: fMRI Evidence in Humans. Brain Stimul. 2015 May-Jun;8(3):624-36. doi: 10.1016/j.brs.2014.11.018. Epub 2014 Dec 6. PMID 25573069
- [Background] Heni M, Wagner R, Kullmann S, Veit R, Mat Husin H, Linder K, Benkendorff C, Peter A, Stefan N, Haring HU, Preissl H, Fritsche A. Central insulin administration improves whole-body insulin sensitivity via hypothalamus and parasympathetic outputs in men. Diabetes. 2014 Dec;63(12):4083-8. doi: 10.2337/db14-0477. Epub 2014 Jul 15. PMID 25028522
- [Result] Gancheva S, Koliaki C, Bierwagen A, Nowotny P, Heni M, Fritsche A, Haring HU, Szendroedi J, Roden M. Effects of intranasal insulin on hepatic fat accumulation and energy metabolism in humans. Diabetes. 2015 Jun;64(6):1966-75. doi: 10.2337/db14-0892. Epub 2015 Jan 9. PMID 25576060